CLINICAL TRIAL: NCT02278939
Title: Filipinos Fit and Trim Weight Loss for Diabetes Prevention Program
Brief Title: Fit and Trim for Diabetes Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Melinda Bender, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-13100; 1R34DK102100-01 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Pre-diabetes; Overweight; Obese
Keywords: diabetes prevention; Filipinos; lifestyle intervention
MeSH Terms: conditions — Glucose Intolerance; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fit and Trim group (Experimental): This groups will start with the Filipinos Fit and Trim Weight Loss Program mobile phone based (smartphone) intervention with social networking for 3 months, a pedometer/accelerometer, access to a study private Facebook virtual social networking group, and and 4 in-person intervention session with individually tailored goals for physical activity, diet, and weight. At 3months, the Fit and Trim group will transition to a maintenance phase for 3 months, receive one in-person session for maintenance support (at 4.5 months) and complete the study at month 6.
  Interventions: Behavioral: Filipinos Fit and Trim Weight Loss Program
- Pedometer only group (Active Comparator): This group will start with the pedometer/accelerometer only to monitor/ track their physical activity step-counts for the initial 3 months. In addition, subjects will receive an educational materials on Hepatitis B and Tuberculosis. At 3 months the pedometer only group will transition to receive the Filipinos Fit and Trim Weight Loss Program intervention (as previously described) for the next 3 months and complete the study at month 6.
  Interventions: Behavioral: Filipinos Fit and Trim Weight Loss Program

INTERVENTIONS:
Behavioral: Filipinos Fit and Trim Weight Loss Program — This 3-month pilot RCT with wait-list control Fit and Trim lifestyle intervention is designed to reduce weight by increasing physical activity, and health eating to improve fasting glucose and hemoglobin A1c. This intervention will use a mobile phone health app diary to self-monitor weight, physical activity, and diet to improve health outcomes to reduce type 2 diabetes risks in Filipino Americans. Program goals are to lose 5% body weight, increase and maintain steps to 12,000 steps/day (20% increase in step-counts each week), reduce total daily fat intake (25% of total calories from fat), and sugar-sweetened beverages over 3 months.
  Other Names: Fit and Trim

SUMMARY:
Filipino Americans (FA) are the second largest (3.4 million) Asian group in the US. and have one of the highest prevalences of obesity and type 2 diabetes mellitus compared to non-Hispanic whites, African Americans and Hispanics. However, FA have been underrepresented in health related research, particularly in diabetes prevention. This proposed pilot study is the first clinical trial to assess preliminary estimates of the short-term effect of the novel social networking diabetes prevention program lifestyle intervention for this high-risk population.

DETAILED DESCRIPTION:
Filipino Americans (FA) are the second largest (3.4 million) Asian group in the US, and the largest (1.5 million) in California, and have the highest prevalence of obesity and type 2 diabetes mellitus (T2DM) compared to non-Hispanic whites, African Americans and Hispanics. However, there has been little health related research among FA. Improving physical activity (PA) and diet can prevent or delay T2DM, as evidenced by the Diabetes Prevention Program (DPP) lifestyle intervention, resulting in reducing T2DM risks. However, implementing the DPP has been expensive and labor intensive. A more cost-effective approach may be the use of mobile technologies coupled with social networking. Filipinos (95%) are avid mobile phone users and the leading Facebook users. Thus, we propose to test a culturally competent mobile phone-based Diabetes Prevention Program lifestyle and social networking (in-person and virtual) intervention in a pilot 3-month randomized controlled trial (RCT) with a wait list active control design for 50 overweight FA at risk for developing type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:: 1) BMI for Asians > 23 kg/m2, 2) Age > 24 years, 3) Diabetes risk test score52 > 5 points, fasting plasma glucose test between 100 - 125 mg/dl, HbA1c > 5.6% or oral glucose tolerance test (OGTT) between 140-200 mg/dl, 4) physically inactive based on Brief Physical Activity Recall Questionnaire,53 5) no cognitive impairment based on the Mini-Cog test,54 and 7) English speaking. Only one member per household will be allowed to enroll in the study. A smart phone will be provided if necessary.

-

Exclusion Criteria:1) Physician diagnosed diabetes and confirmed by clinical data (e.g. documentation of fasting blood glucose >126 mg/dL or a positive OGTT), 2) HbA1C > 7.0%, 3) Glucose metabolism associated disease (Cushing's syndrome, Acromegaly, and Pheochromocytoma currently under treatment, chronic pancreatitis), 4) Thyroid disease - sub-optimally treated, 5) Known medical conditions or other physical problems needing special exercise program (e.g., prior myocardial infarction, history of angioplasty or angina, admission for hospital evaluation of chest pain, use of nitroglycerin for angina, asthma, chronic obstructive pulmonary disease, or uncontrolled hypertension), 6) Currently participating in a lifestyle modification program, 7) Planning a trip outside of the US during the 3-month study period, 8) Known eating disorder, 9) Planning to have gastric bypass surgery, 10) Taking antibiotics (including HIV-related agents), anti-tuberculosis agents (except tuberculosis prophylaxis)], or prescription weight-loss drugs.

-

Ages: 24 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda S Bender, PhD, RN, Principal Investigator — University of California, San Francisco; Yoshimi Fukuoka, PhD, RN, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco / Daly City Communities, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated under this project will be administered in accordance with both University and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance of March 5, 2003. That data set will be made available to qualified investigators within one year after completion of our investigators' data analyses and publication of papers presenting the results of those analyses.
  Requests will be reviewed and acted on by the PI or in consultation with a UCSF representative. After approval, the PI will prepare the requested dataset. This dataset will be carefully screened to make certain that all identifying information has been removed, including information that could be combined so as to identify an individual. Data will be provided in comma separated variables (CSV) text format rather than a proprietary format either on a CD or through a password-protected download from our website.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: That data set will be made available to qualified investigators within one year after completion of our investigators' data analyses and publication of papers presenting the results of those analyses.
Access Criteria: Data generated under this project will be administered in accordance with both University and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance of March 5, 2003. Requests will be reviewed and acted on by the PI or in consultation with a UCSF representative. After approval, the PI will prepare the requested dataset. This dataset will be carefully screened to make certain that all identifying information has been removed, including information that could be combined so as to identify an individual. Data will be provided in comma separated variables (CSV) text format rather than a proprietary format either on a CD or through a password-protected download from our website.

REFERENCES:
- [Derived] Chang L, Fukuoka Y, Aouizerat BE, Zhang L, Flowers E. Prediction of Weight Loss to Decrease the Risk for Type 2 Diabetes Using Multidimensional Data in Filipino Americans: Secondary Analysis. JMIR Diabetes. 2023 Apr 11;8:e44018. doi: 10.2196/44018. PMID 37040172
- [Derived] Bender MS, Cooper BA, Flowers E, Ma R, Arai S. Filipinos Fit and Trim - A feasible and efficacious DPP-based intervention trial. Contemp Clin Trials Commun. 2018 Sep 20;12:76-84. doi: 10.1016/j.conctc.2018.09.004. eCollection 2018 Dec. PMID 30294699

RESULTS

PARTICIPANT FLOW:
Groups:
- Fit and Trim Group: This groups will start with the Filipinos Fit and Trim Weight Loss Program mobile phone based (smartphone) intervention with social networking for 3 months, a pedometer/accelerometer, access to a study private Facebook virtual social networking group, and and 4 in-person intervention session with individually tailored goals for physical activity, diet, and weight. At 3months, the Fit and Trim group will transition to a maintenance phase for 3 months, receive one in-person session for maintenance support (at 4.5 months) and complete the study at month 6.
  Filipinos Fit and Trim Weight Loss Program: This 3-month pilot RCT with wait-list control Fit and Trim lifestyle intervention is designed to reduce weight by increasing physical activity, and health eating to improve fasting glucose and hemoglobin A1c. This intervention uses a mobile phone health app diary to self-monitor weight, physical activity, and diet to improve health outcomes to reduce type 2 diabetes risks in Filipino
- Pedometer Only Group: This group will start with the pedometer/accelerometer only to monitor/ track their physical activity step-counts for the initial 3 months. In addition, subjects will receive an educational materials on Hepatitis B and Tuberculosis. At 3 months pedometer only group will transition to receive the Filipinos Fit and Trim Weight Loss Program intervention (as previously described) for the next 3 months and complete the study at month 6.
  Filipinos Fit and Trim Weight Loss Program: This 3-month pilot RCT with wait-list control Fit and Trim lifestyle intervention is designed to reduce weight by increasing physical activity, and health eating to improve fasting glucose and hemoglobin A1c. This intervention will use a mobile phone health app diary to self-monitor weight, physical activity, and diet to improve health outcomes to reduce type 2 diabetes risks in Filipino Americans. Program goals are to lose 5% body weight, increase and maintain steps to 12,000 steps/day (20% increase in st
Period: Overall Study
Arm/Group | Fit and Trim Group | Pedometer Only Group
Started | 33 | 34
Completed | 28 | 33
Not Completed | 5 | 1
Not completed — lack of time | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — death in family | 1 | 0
Not completed — family emergency unable to commit | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fit and Trim Group | Pedometer Only Group | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (12.1) | 42.1 (12.1) | 41.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 17 | 15 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 34 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 33 | 34 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 00 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Who Completed the Study
Description: at least 85% of participants enrolled complete the study program
Time Frame: Baseline to 6-months
Population: Eligible participants enrolled and randomized = 67 ( Intervention group = 33 Control group =34). A Feasibility = at least 85% of all enrolled participant will have completed the study program.
Measure: Count of Participants; unit: Participants
Groups:
- Fit and Trim Intervention Group: This groups immediately starts the Filipinos Fit and Trim Weight Loss Program mobile phone based (smartphone) intervention with social networking for the initial 3 months. At 3months, the Fit and Trim group transitions to a 3-month maintenance phase and completes the study at the 6-month visit.
  Filipinos Fit and Trim Weight Loss Program: This 3-month pilot RCT with wait-list control Fit and Trim lifestyle intervention is designed to reduce weight by increasing physical activity, and health eating to improve fasting glucose and hemoglobin A1c. This intervention will use a mobile phone health app diary to self-monitor weight, physical activity, and diet to improve health outcomes to reduce type 2 diabetes risks in Filipino Americans. Program goals are to lose 5% body weight, increase and maintain steps to 12,000 steps/day (20% increase in step-counts each week), reduce total daily fat intake (25% of total calories from fat), and sugar-sweetened beverages over 3 months.
- Active Control Group: This group starts using the Fitbit accelerometer only to track physical activity step-counts for the initial 3 months. At the 3 month visit, the active control participants transition to receive the 3-month Filipinos Fit and Trim intervention and complete the study at their 6-month visit.
  Filipinos Fit and Trim Weight Loss Program: This 3-month pilot RCT with wait-list control Fit and Trim lifestyle intervention is designed to reduce weight by increasing physical activity, and health eating to improve fasting glucose and hemoglobin A1c. This intervention will use a mobile phone health app diary to self-monitor weight, physical activity, and diet to improve health outcomes to reduce type 2 diabetes risks in Filipino Americans. Program goals are to lose 5% body weight, increase and maintain steps to 12,000 steps/day (20% increase in step-counts each week), reduce total daily fat intake (25% of total calories from fat), and sugar-sweetened beverages over 3 months.
Arm/Group | Fit and Trim Intervention Group | Active Control Group
Number analyzed (Participants) | 33 | 34
Participants | 28 | 33

2. Secondary Outcome: Weight Change in Kilogram
Description: Weight change in kilogram by group
Time Frame: Baseline to 3 months
Population: Overweight/obese English-speaking Filipino American adults were randomized in a 1:1 ratio either to the intervention group or active control group.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Fit and Trim Intervention Group | Active Control Group
Number analyzed (Participants) | 28 | 33
kilograms | -3.4 (3.6) | -0.9 (2.5)
Statistical Analysis 1: Comparison: Fit and Trim Intervention Group vs Active Control Group; Hypothesis: the intervention group will have a significantly greater reduction in weight (kg) compared to the control from baseline to 3-months; Test type: Superiority; p = 0.003, ANOVA — This was an intention to treat analysis using the Tukey-Kramer adjustment to account for unequal group sample sizes

3. Secondary Outcome: Percent of Weight
Description: Percent of weight change from baseline to 3-months by group
Time Frame: Baseline to 3 months
Population: Overweight/obese English-speaking Filipino American adults were randomized either to the Intervention group or the active control.
Measure: Mean (Standard Deviation); unit: percent of weight
Arm/Group | Fit and Trim Intervention Group | Active Control Group
Number analyzed (Participants) | 28 | 33
percent of weight | -4.33 (4.26) | -1.02 (3.14)
Statistical Analysis 1: Comparison: Fit and Trim Intervention Group vs Active Control Group; Hypothesis: the intervention group will have a statistically greater reduction in percent weight compared to the control from baseline to 3-months; Test type: Superiority; p = .001, ANOVA — This was an intention to treat analysis using the Tukey-Kramer adjustment to account for unequal group sample sizes

4. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in body mass index per group
Time Frame: Baseline to 3 months
Population: Overweight/obese English-speaking Filipino American adults, were randomized either to the Intervention group (received a combination of mobile app, social media and in-person diabetes prevention intervention) or the active control group.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Fit and Trim Intervention Group | Active Control Group
Number analyzed (Participants) | 28 | 33
kg/m^2 | -1.27 (1.29) | -0.33 (.95)
Statistical Analysis 1: Comparison: Fit and Trim Intervention Group vs Active Control Group; Hypothesis: the intervention group will have a statistically greater reduction in BMI compared to the control from baseline to 3 months; Test type: Superiority; p = .002, ANOVA — This was an intention to treat analysis using the Tukey-Kramer adjustment to account for differences in group sample sizes

ADVERSE EVENTS:
Time Frame: 1.5 years (Dec 2014 through June 2016)
Description: This study complied with the same clinicaltrials.gov definition for adverse event and/or serious adverse event. At each participant's scheduled research office visit an adverse event questionnaire was completed by the research staff to assess if any participant adverse events and/or serious adverse event had occurred since the previous research office visit.
Groups:
- Fit and Trim Group: This groups immediately starts Filipinos Fit and Trim Weight Loss Program mobile phone intervention with social networking for the first 3 months, At 3months, the Fit and Trim group transitions to a maintenance phase for another 3 months, and completes the study at month 6.
  Filipinos Fit and Trim Weight Loss Program: This 3-month pilot RCT with wait-list control Fit and Trim lifestyle intervention is designed to reduce weight by increasing physical activity, and health eating to improve fasting glucose and hemoglobin A1c. This intervention will use a mobile phone health app diary to self-monitor weight, physical activity, and diet to improve health outcomes to reduce type 2 diabetes risks in Filipino Americans. Program goals are to lose 5% body weight, increase and maintain steps to 12,000 steps/day (20% increase in step-counts each week), reduce total daily fat intake (25% of total calories from fat), and sugar-sweetened beverages over 3 months.
- Pedometer Only Group: This group starts with a Fitbit pedometer/accelerometer only for the initial 3 months. At 3 months the pedometer only group transitions to receive the Filipinos Fit and Trim Weight Loss Program intervention ) for the next 3 months and completes the study at month 6.
  Filipinos Fit and Trim Weight Loss Program: This 3-month pilot RCT with wait-list control Fit and Trim lifestyle intervention is designed to reduce weight by increasing physical activity, and health eating to improve fasting glucose and hemoglobin A1c. This intervention will use a mobile phone health app diary to self-monitor weight, physical activity, and diet to improve health outcomes to reduce type 2 diabetes risks in Filipino Americans. Program goals are to lose 5% body weight, increase and maintain steps to 12,000 steps/day (20% increase in step-counts each week), reduce total daily fat intake (25% of total calories from fat), and sugar-sweetened beverages over 3 months.
Arm/Group | Fit and Trim Group | Pedometer Only Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34

LIMITATIONS AND CAVEATS:
Due to the overall small sample size (n=67) and recruitment restricted to one geographical region, study results cannot be generalized to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No